CLINICAL TRIAL: NCT03112135
Title: Effect of Topical and Systemic Tranexemic Acid on Bleeding and Quality of Surgical Field During Ear Exploration Surgery. A Double Blind Randomized Clinical Trial
Brief Title: Effect of Topical and Systemic Tranexemic Acid on Bleeding During Ear Exploration Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sally Ahmed kamel, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: assuit university hospital
Record Dates: First submitted 2017-03-06; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Intraoperative Bleeding
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Systemic TXA (Active Comparator): TXA 10-15 mg i.v over 30 min. followed by infusion in a dose of 1 mg / kg /hr
  Interventions: Drug: Tranexamic Acid
- Topical TXA (Active Comparator): Topical TXA 1 gm diluted in 200 ml saline
  Interventions: Drug: Tranexamic Acid
- Topical adrenaline (Active Comparator): Topical adrenaline 1 mg diluted in 200 ml saline
  Interventions: Drug: Adrenalin

INTERVENTIONS:
Drug: Tranexamic Acid — TXA of 10-15 mg i.v over 30 min. followed by infusion in adose of 1 mg / kg /hr
  Other Names: kapron
  Arms: Systemic TXA
Drug: Tranexamic Acid — Topical TXA 1 gm diluted in 200 ml saline
  Other Names: kapron
  Arms: Topical TXA
Drug: Adrenalin — Topical adrenaline 1 mg diluted on 200 ml saline
  Other Names: Epinephrine
  Arms: Topical adrenaline

SUMMARY:
The effect of tranexamic acid (TXA) on bleeding and improvement of surgical field during ear exploration surgery is not clear yet. This study will conducted to answer this question.

DETAILED DESCRIPTION:
Bleeding during ear surgery is still a challenge for surgeons and anesthesiologists . Although extensive blood loss is rare during ear surgery, however, establishing a favorite surgical field is often difficult. The reason is that even slight bleeding may distort the view of the field and increase the occurrence of complications, including deafness, the longer duration of surgery, or even inconclusive surgery .

Many techniques have been proposed to improve the field of ear exploration surgery. Bipolar diathermy, packing, local vasoconstrictors, and induced hypotension are the most commonly used techniques . Diathermy can lead to local damage and delayed bleeding . Using topical vasoconstrictions can lead to hemodynamic instability especially in patients with a history of hypertension or ischemic heart disease. Induction hypotension exposes the patients to more anesthetic drugs and hence a higher risk of potential side effects. However, neither of these methods guarantees a desirable surgical field with no bleeding. Therefore, investigators are working on more effective and safer methods to reduce bleeding and hence to improve the field of surgery .

Activation of fibrinolysis during and after surgery is a well-known phenomenon. Many mechanisms associated with coagulation disorders, such as surgical trauma, blood loss and consumption of coagulation factors and platelets, using crystalloid and colloid given during and after surgery, hypothermia, acidosis, foreign materials, and etc. In recent studies, systemic infusion of anti-fibrinolytic drugs have been used to reduce bleeding in various forms of surgery such as major orthopedic surgery,and adeno-tonsillectomy.

Tranexamic acid (TXA) is a synthetic antifibrinolytic agent that binds to the lysine binding sites of plasmin and plasminogen. Saturation of the binding sites causes separation of plasminogen from superficial fibrin and hence prevents fibrinolysis. Any surgical procedure can cause a considerable tissue damage and hence trigger the release of enzymes, such as 'tissue plasminogen activator' that converts plasminogen to plasmin and activates fibrinolysis process. TXA can prevent fibrinolysis activity by inhibiting the activity of this enzyme.

Systemic infusion of TXA associated with several potential side effects such as nausea, vomiting, diarrhea, allergic dermatitis, dizziness, hypotension, seizures, impaired vision, achromatopsia (impaired color vision), and particularly thromboembolic events. Several studies have been conducted on topical TXA in different types of surgery but no systemic absorption or side effects have been reported.

To date, the effect of TXA on reduction of bleeding in ear surgery is unclear . There is no consensus on the efficacy of TXA and its effective dose in reducing bleeding. This trial will aim to assess the effect of topical TXA on bleeding and improvement of surgical field during ear surgery in patients with chronic ear disease.

ELIGIBILITY:
Inclusion Criteria:

1. being candidate for ear exploration surgery.
2. ASA I-II
3. Willing to participate in the study
4. Hb level > 10 mg/dl.
5. normal coagulation profile (INR and PTT )

Exclusion Criteria:

1. Patient refusal
2. allergy toTXA
3. Bleeding disorder
4. psychiatric illness
5. acute and chronic renal failure
6. using heparin during 48 hr before surgery
7. pregnancy
8. cirrhosis
9. colour blindness
10. cardiac stent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The quality of the surgical field | 45 minutes after the start of surgery
  Boezaart grading with 0-5 scores.

SECONDARY OUTCOMES:
intraoperative blood loss | 45 minutes after the start of surgery
  Blood in the suction and the gauze

CONTACTS AND LOCATIONS:
Overall Officials: Sally Ahmed, Dr, Principal Investigator — Assiut Univerisity
Locations (1):
- Egypt, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No